CLINICAL TRIAL: NCT01594515
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 1015550 in Healthy Male Volunteers (a Partially Randomised, Partially Single-blind, Placebo-controlled Phase I Study)
Brief Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 1015550 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1305.1; 2012-000405-68 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550

ARMS (10):
- BI 1015550 low dose A (Experimental): Powder for oral solution
  Interventions: Drug: BI 1015550
- BI 1015550 low dose B (Experimental): Powder for oral solution
  Interventions: Drug: BI 1015550
- BI 1015550 low dose C (Experimental): Powder for oral solution
  Interventions: Drug: BI 1015550
- BI 1015550 low dose D (Experimental): Powder for oral solution
  Interventions: Drug: BI 1015550
- BI 1015550 medium dose A (Experimental): Powder for oral solution
  Interventions: Drug: BI 1015550
- BI 1015550 medium dose B (Experimental): Powder for oral solution
  Interventions: Drug: BI 1015550
- BI 1015550 medium dose C (Experimental): Powder for oral solution
  Interventions: Drug: BI 1015550
- BI 1015550 high dose A (Experimental): Powder for oral solution
  Interventions: Drug: BI 1015550
- BI 1015550 high dose B (Experimental): Powder for oral solution
  Interventions: Drug: BI 101550
- Placebo (Placebo Comparator): Solution for oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1015550 — High dose powder for oral solution
  Arms: BI 1015550 high dose A
Drug: BI 1015550 — Medium dose powder for oral solution
  Arms: BI 1015550 medium dose A
Drug: BI 1015550 — Low dose powder for oral solution
  Arms: BI 1015550 low dose C
Drug: BI 1015550 — Low dose powder for oral solution
  Arms: BI 1015550 low dose B
Drug: BI 1015550 — Low dose powder for oral solution
  Arms: BI 1015550 low dose A
Drug: Placebo — Solution for oral administration
  Arms: Placebo
Drug: BI 101550 — High dose powder for oral solution
  Arms: BI 1015550 high dose B
Drug: BI 1015550 — Low dose powder for oral solution
  Arms: BI 1015550 low dose D
Drug: BI 1015550 — Medium dose powder for oral solution
  Arms: BI 1015550 medium dose C
Drug: BI 1015550 — Medium dose powder for oral solution
  Arms: BI 1015550 medium dose B

SUMMARY:
In this first-in-man trial, safety, tolerability, pharmacokinetics, and selected pharmacodynamics parameters of BI 1015550 will be assessed in healthy male volunteers.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1305.1.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 patients were treated and analysed.
Pre-assignment Details: Partially randomised, placebo-controlled within dose groups, single-blinded, single-centre study to assess the safety, tolerability and pk of single rising oral doses of BI 1015550(a powder for oral solution reconstituted with solvent tartaric acid and solvent component hydroxy-propyl-β-cyclodextrin (HPβCD)) in healthy male volunteers.
Groups:
- BI 1015550 Low Dose 0.02mg: Single oral dose of 0.02mg powder solution of BI 1015550 were administered once a day after an overnight fast to healthy male volunteers.
- BI 1015550 Low Dose 0.06mg: Single oral dose of 0.06mg powder solution of BI 1015550 were administered once a day after an overnight fast to healthy male volunteers.
- BI 1015550 Low Dose 0.2mg: Single oral dose of 0.2mg powder solution of BI 1015550 were administered once a day after an overnight fast to healthy male volunteers.
- BI 1015550 Low Dose 0.6mg: Single oral dose of 0.6mg powder solution of BI 1015550 were administered once a day after an overnight fast to healthy male volunteers.
- BI 1015550 Medium Dose 2mg: Single oral dose of 2mg powder solution of BI 1015550 were administered once a day after an overnight fast to healthy male volunteers.
- BI 1015550 Medium Dose 4mg: Single oral dose of 4mg powder solution of BI 1015550 were administered once a day after an overnight fast to healthy male volunteers.
- BI 1015550 Medium Dose 8mg: Single oral dose of 8mg powder solution of BI 1015550 were administered once a day after an overnight fast to healthy male volunteers.
- BI 1015550 High Dose 16mg: Single oral dose of 16mg powder solution of BI 1015550 were administered once a day after an overnight fast to healthy male volunteers.
- BI 1015550 High Dose 24mg: Single oral dose of 24mg powder solution of BI 1015550 were administered once a day after an overnight fast to healthy male volunteers.
- Placebo: Single oral dose of placebo powder solution with matching volume were administered once a day after an overnight fast to healthy male volunteers.
Period: Overall Study
Arm/Group | BI 1015550 Low Dose 0.02mg | BI 1015550 Low Dose 0.06mg | BI 1015550 Low Dose 0.2mg | BI 1015550 Low Dose 0.6mg | BI 1015550 Medium Dose 2mg | BI 1015550 Medium Dose 4mg | BI 1015550 Medium Dose 8mg | BI 1015550 High Dose 16mg | BI 1015550 High Dose 24mg | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The treated set (TS) included all subjects who were dispensed study medication and were documented to have taken at least 1 dose of the investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1015550 Low Dose 0.02mg | BI 1015550 Low Dose 0.06mg | BI 1015550 Low Dose 0.2mg | BI 1015550 Low Dose 0.6mg | BI 1015550 Medium Dose 2mg | BI 1015550 Medium Dose 4mg | BI 1015550 Medium Dose 8mg | BI 1015550 High Dose 16mg | BI 1015550 High Dose 24mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.5 (5.1) | 29.5 (4.8) | 38.2 (6.5) | 35.0 (5.5) | 35.5 (5.9) | 32.7 (5.9) | 36.3 (6.3) | 40.5 (3.3) | 33.5 (8.4) | 36.6 (5.6) | 35.3 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number (%) of Subjects With Drug Related Adverse Events
Description: Percentage of subjects with drug related adverse events.
Time Frame: From the day of informed consent(-21 days) until the end-of-study examination(within 5 to 7 days after last PK sampling), upto 10 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | BI 1015550 Low Dose 0.02mg | BI 1015550 Low Dose 0.06mg | BI 1015550 Low Dose 0.2mg | BI 1015550 Low Dose 0.6mg | BI 1015550 Medium Dose 2mg | BI 1015550 Medium Dose 4mg | BI 1015550 Medium Dose 8mg | BI 1015550 High Dose 16mg | BI 1015550 High Dose 24mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Percentage of Participants | 0.0 | 33.3 | 16.7 | 0.0 | 0.0 | 33.3 | 16.7 | 16.7 | 16.7 | 6.3

2. Primary Outcome: Number (%) of Subjects With Clinically Relevant Abnormalities in Clinical Laboratory Tests
Description: Percentage of subjects with clinically relevant abnormalities in clinical laboratory tests (haematology, clinical chemistry, haemoccult® test, and urinalysis).
Time Frame: Day -21 to -2, upto -72 hours, 4h, 24h, 48h, 72h and study examination(within 5 to 7 days after last PK sampling).
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | BI 1015550 Low Dose 0.02mg | BI 1015550 Low Dose 0.06mg | BI 1015550 Low Dose 0.2mg | BI 1015550 Low Dose 0.6mg | BI 1015550 Medium Dose 2mg | BI 1015550 Medium Dose 4mg | BI 1015550 Medium Dose 8mg | BI 1015550 High Dose 16mg | BI 1015550 High Dose 24mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

3. Primary Outcome: Number (%) of Subjects With Clinically Relevant Abnormalities in Vital Signs
Description: Percentage of subjects with clinically relevant abnormalities in vital signs (blood pressure, pulse rate, respiratory rate, oral body temperature, orthostasis test).
Time Frame: Day -21 to -2, -1 hour, 0.5h, 1h, 2h, 4h, 8h, 10h, 24h, 48h, 72h and study examination(within 5 to 7 days after last PK sampling).
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | BI 1015550 Low Dose 0.02mg | BI 1015550 Low Dose 0.06mg | BI 1015550 Low Dose 0.2mg | BI 1015550 Low Dose 0.6mg | BI 1015550 Medium Dose 2mg | BI 1015550 Medium Dose 4mg | BI 1015550 Medium Dose 8mg | BI 1015550 High Dose 16mg | BI 1015550 High Dose 24mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

4. Primary Outcome: Number (%) of Subjects With Clinically Relevant Abnormalities in 12-lead ECGs
Description: Percentage of subjects with clinically relevant abnormalities in 12-lead ECGs.
Time Frame: as for outcome 3
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | BI 1015550 Low Dose 0.02mg | BI 1015550 Low Dose 0.06mg | BI 1015550 Low Dose 0.2mg | BI 1015550 Low Dose 0.6mg | BI 1015550 Medium Dose 2mg | BI 1015550 Medium Dose 4mg | BI 1015550 Medium Dose 8mg | BI 1015550 High Dose 16mg | BI 1015550 High Dose 24mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

5. Primary Outcome: Number (%) of Subjects With Clinically Relevant Abnormalities in Tolerability
Description: Percentage of subjects with clinically relevant abnormalities in tolerability assessed by the investigator.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | BI 1015550 Low Dose 0.02mg | BI 1015550 Low Dose 0.06mg | BI 1015550 Low Dose 0.2mg | BI 1015550 Low Dose 0.6mg | BI 1015550 Medium Dose 2mg | BI 1015550 Medium Dose 4mg | BI 1015550 Medium Dose 8mg | BI 1015550 High Dose 16mg | BI 1015550 High Dose 24mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

6. Primary Outcome: Number (%) of Subjects With Clinically Relevant Abnormalities in Physical Examinations
Description: Percentage of subjects with clinically relevant abnormalities in physical examinations.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | BI 1015550 Low Dose 0.02mg | BI 1015550 Low Dose 0.06mg | BI 1015550 Low Dose 0.2mg | BI 1015550 Low Dose 0.6mg | BI 1015550 Medium Dose 2mg | BI 1015550 Medium Dose 4mg | BI 1015550 Medium Dose 8mg | BI 1015550 High Dose 16mg | BI 1015550 High Dose 24mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

7. Secondary Outcome: Cmax of BI 1015550
Description: Maximum measured concentration of the analyte in plasma.
Time Frame: -0.5hour before dosing and 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after dosing
Population: The pharmacokinetic analysis set (PKS) included all subjects in the TS who provided at least 1 evaluable observation for a PK endpoint. A subject was considered to be evaluable if he provided sufficient data, did not vomit at or before 2x median tmax and completed the trial without any iPV relevant to the PK evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | BI 1015550 Low Dose 0.02mg | BI 1015550 Low Dose 0.06mg | BI 1015550 Low Dose 0.2mg | BI 1015550 Low Dose 0.6mg | BI 1015550 Medium Dose 2mg | BI 1015550 Medium Dose 4mg | BI 1015550 Medium Dose 8mg | BI 1015550 High Dose 16mg | BI 1015550 High Dose 24mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nmol/L | NA (NA) — Not calculated because BI 1015550 was below the detection limit | 1.42 (23.2) | 5.02 (20.1) | 13.7 (14.2) | 46.9 (38.9) | 113 (20.4) | 176 (12.6) | 292 (22.2) | 542 (12.1)
Statistical Analysis 1: Comparison: BI 1015550 Low Dose 0.06mg vs BI 1015550 Low Dose 0.2mg vs BI 1015550 Low Dose 0.6mg vs BI 1015550 Medium Dose 2mg vs BI 1015550 Medium Dose 4mg vs BI 1015550 Medium Dose 8mg vs BI 1015550 High Dose 16mg vs BI 1015550 High Dose 24mg; This was non confirmatory testing (Single dose). Dose proportionality of the drug for Cmax was analysed.(N=50); Test type: Superiority or Other; Slope = 0.9702, 95% CI 2-sided [0.9400 to 1.0005], Standard Error of Mean 0.0151 — Dose proportionality was explored using the power model (ANCOVA). The perfect dose proportionality would correspond to a slope β of 1. PK endpoints on the log-transformed scale

8. Secondary Outcome: AUC0-infinity of BI 1015550
Description: Area under the concentration-time curve in plasma over the time interval from 0 extrapolated to infinity
Time Frame: -0.5hour before dosing and 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after dosing
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 1015550 Low Dose 0.02mg | BI 1015550 Low Dose 0.06mg | BI 1015550 Low Dose 0.2mg | BI 1015550 Low Dose 0.6mg | BI 1015550 Medium Dose 2mg | BI 1015550 Medium Dose 4mg | BI 1015550 Medium Dose 8mg | BI 1015550 High Dose 16mg | BI 1015550 High Dose 24mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nmol*h/L | NA (NA) — Not calculated because BI 1015550 was below the detection limit | 7.44 (12.7) | 24.1 (13.9) | 67.9 (15.6) | 287 (14.9) | 679 (32.0) | 1210 (18.3) | 2180 (19.9) | 3650 (22.6)
Statistical Analysis 1: Comparison: BI 1015550 Low Dose 0.06mg vs BI 1015550 Low Dose 0.2mg vs BI 1015550 Low Dose 0.6mg vs BI 1015550 Medium Dose 2mg vs BI 1015550 Medium Dose 4mg vs BI 1015550 Medium Dose 8mg vs BI 1015550 High Dose 16mg vs BI 1015550 High Dose 24mg; This was non confirmatory testing (Single dose). Dose proportionality of the drug for AUC0-inf was analysed. (N=48); Test type: Superiority or Other; Slope = 1.0442, 95% CI 2-sided [1.0145 to 1.0740], Standard Error of Mean 0.0148 — [estimate comment as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: From the day of informed consent(-21 days) until the end-of-study examination(within 5 to 7 days after last PK sampling), upto 10 days.
Arm/Group | Placebo | BI 1015550 Low Dose 0.02mg | BI 1015550 Low Dose 0.06mg | BI 1015550 Low Dose 0.2mg | BI 1015550 Low Dose 0.6mg | BI 1015550 Medium Dose 2mg | BI 1015550 Medium Dose 4mg | BI 1015550 Medium Dose 8mg | BI 1015550 High Dose 16mg | BI 1015550 High Dose 24mg
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/16 | 2/6 | 2/6 | 3/6 | 3/6 | 1/6 | 3/6 | 3/6 | 2/6 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | BI 1015550 Low Dose 0.02mg (N=6) | BI 1015550 Low Dose 0.06mg (N=6) | BI 1015550 Low Dose 0.2mg (N=6) | BI 1015550 Low Dose 0.6mg (N=6) | BI 1015550 Medium Dose 2mg (N=6) | BI 1015550 Medium Dose 4mg (N=6) | BI 1015550 Medium Dose 8mg (N=6) | BI 1015550 High Dose 16mg (N=6) | BI 1015550 High Dose 24mg (N=6)
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
BI 1015550 high dose 24mg was originally planned as 26 mg but reduced due to PK interim analysis results of previous dose group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No